CLINICAL TRIAL: NCT02783729
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Active Comparator, Parallel-Group Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older With Insomnia Disorder (SUNRISE 1)
Brief Title: Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older With Insomnia Disorder (SUNRISE 1)
Acronym: SUNRISE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-G000-304; 2015-004347-39 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2018-03

CONDITIONS: Insomnia
Keywords: E2006; Lemborexant; zolpidem tartrate; Ambien CR; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Lemborexant 5 milligrams (mg) (Experimental): Participants will receive one lemborexant 5 mg tablet and one zolpidem-matched placebo tablet each night
  Interventions: Drug: Lemborexant; Drug: Zolpidem-matched placebo
- Lemborexant 10 mg (Experimental): Participants will receive one lemborexant 10 mg tablet and one zolpidem-matched placebo tablet each night
  Interventions: Drug: Lemborexant; Drug: Zolpidem-matched placebo
- Zolpidem tartrate (Active Comparator): Participants will receive one zolpidem 6.25 mg tablet and one lemborexant-matched placebo tablet each night
  Interventions: Drug: Lemborexant-matched placebo; Drug: Zolpidem tartrate
- Placebo (Placebo Comparator): Participants will receive one zolpidem-matched placebo tablet and one lemborexant-matched placebo tablet each night
  Interventions: Drug: Lemborexant-matched placebo; Drug: Zolpidem-matched placebo

INTERVENTIONS:
Drug: Lemborexant — Lemborexant 5 mg will be administered orally in tablet form at home each night, immediately before the time the participant intends to try to sleep.
  Other Names: E2006
  Arms: Lemborexant 5 milligrams (mg)
Drug: Lemborexant — Lemborexant 10 mg will be administered orally in tablet form at home each night, immediately before the time the participant intends to try to sleep.
  Other Names: E2006
  Arms: Lemborexant 10 mg
Drug: Lemborexant-matched placebo — Lemborexant-matched placebo be administered orally in tablet form at home each night, immediately before the time the participant intends to try to sleep.
  Arms: Placebo; Zolpidem tartrate
Drug: Zolpidem tartrate — Zolpidem tartrate extended release 6.25 mg will be administered orally in tablet form at home each night, immediately before the time the participant intends to try to sleep.
  Other Names: Ambien CR
  Arms: Zolpidem tartrate
Drug: Zolpidem-matched placebo — Zolpidem-matched placebo will be administered orally in tablet form at home each night, immediately before the time the participant intends to try to sleep.
  Arms: Lemborexant 10 mg; Lemborexant 5 milligrams (mg); Placebo

SUMMARY:
This study will be conducted to demonstrate, using polysomnography, that lemborexant 10 milligrams (mg) and 5 mg is superior to placebo on objective sleep onset as assessed by latency to persistent to sleep (LPS) after the last 2 nights of 1 month of treatment in participants 55 years and older with insomnia disorder.

DETAILED DESCRIPTION:
The study is a multicenter, randomized, double-blind, placebo-controlled, active comparator, parallel-group study of 2 dose levels of lemborexant for 30 nights in approximately 950 participants, 55 years or older with insomnia disorder. Participants will be males 65 years or older or females 55 years or older. Approximately 60% of the participants will be age 65 years or older. The study will have 2 phases: The Prerandomization Phase and the Randomization Phase. Including both phases, the study will last for a minimum of 65 and a maximum of 81 days per participant.

ELIGIBILITY:
Inclusion Criteria

1. Male age 65 years or older or female age 55 years or older at the time of informed consent
2. Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for Insomnia Disorder, as follows:

   * Complains of dissatisfaction with nighttime sleep, in the form of difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep (Note that if the complaint is limited to difficulty initiating sleep, the participant is not eligible)
   * Frequency of complaint ≥ 3 times per week
   * Duration of complaint ≥ 3 months
   * Associated with complaint of daytime impairment
3. History of subjective wake after sleep onset (sWASO) typically ≥ 60 minutes on at least 3 nights per week in the previous 4 weeks
4. Reports regular time spent in bed, either sleeping or trying to sleep, between 7 and 9 hours
5. Reports habitual bedtime, defined as the time the participant attempts to sleep, between 21:00 and 24:00 and habitual waketime between 05:00 and 09:00
6. Insomnia Severity Index (ISI) score ≥ 13
7. Confirmation of current insomnia symptoms as determined from responses on the Sleep Diary before the second screening visit
8. Confirmation of regular bedtime and waketime as determined from responses on the Sleep Diary
9. Confirmation of sufficient duration of time spent in bed, as determined from responses on the Sleep Diary
10. Objective (polysomnography [PSG]) evidence of insomnia as follows:

    a) Wake after sleep onset (WASO) average ≥ 60 minutes on the 2 consecutive PSGs, with neither night < 45 minutes
11. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
12. Willing not to start a behavioral or other treatment program for the treatment of insomnia during the participant's participation in the study

Exclusion Criteria

1. A current diagnosis of sleep-related breathing disorder including obstructive sleep apnea (with or without continuous positive airway pressure [CPAP] treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows:

   1. STOPBang score ≥5
   2. International Restless Legs Scale score ≥16
   3. Epworth Sleepiness Scale score >15 (scores of 11 to 15 require excessive daytime sleepiness to be recorded in participant's Medical History)
2. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
3. On the Munich Parasomnia Scale (MUPS), endorsed the item that corresponds to a history of sleep-eating or reports a history of sleep-related violent behavior, sleep-driving, or symptoms of another parasomnia that in the investigator's opinion make the participant unsuitable for the study
4. Apnea-Hypopnea Index > 15 or Periodic Limb Movement with Arousal Index >15 as measured on the PSG at the second screening visit
5. Beck Depression Inventory - II (BDI-II) score >19 at Screening
6. Beck Anxiety Index (BAI) score >15 at Screening
7. Habitually naps during the day more than 3 times per week
8. Is a female of childbearing potential Note: All females will be considered to be of childbearing potential unless they are postmenopausal (defined as amenorrheic for at least 12 consecutive months, and are postmenopausal without other known or suspected cause), or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
9. Excessive caffeine use that in the opinion of the investigator contributes to the participant's insomnia, or habitually consumes caffeine-containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study.
10. History of drug or alcohol dependency or abuse within approximately the previous 2 years
11. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males), or unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
12. Known to be positive for human immunodeficiency virus
13. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
14. A prolonged QT/QTcF interval (QTcF >450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG) at Screening (repeated only if initial ECG indicates a QTcF interval >450 ms)
15. Current evidence of clinically significant disease (e.g., cardiac; respiratory including chronic obstructive pulmonary disease, acute and/or severe respiratory depression; gastrointestinal; severe hepatic impairment; renal including severe renal impairment; neurological including myasthenia gravis; psychiatric disease; or malignancy within the past 5 years other than adequately treated basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments, including the ability to perform tasks on the cognitive performance assessment battery (PAB). Participants for whom a sedating drug would be contraindicated for safety reasons because of the participant's occupation or activities are also excluded.
16. Comorbid nocturia resulting in frequent need to get out of bed to use the bathroom during the night
17. Any history of a medical or psychiatric condition that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessment, including the ability to perform the PAB.
18. Any suicidal ideation with intent with or without a plan, at the time of or within 6 months before the electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) administration during the Prerandomization Phase (i.e., answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the eC-SSRS)
19. Any suicidal behavior in the past 10 years (per the Suicidal Behavior section of the eC-SSRS)
20. Scheduled for surgery during the study
21. Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half lives, whichever is longer, before the first dose of study medication (Run-in Period).
22. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period)
23. Failed treatment with suvorexant (Belsomra®) (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
24. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel across more than 3 time zones during the study
25. A positive drug test at Screening, Run-In, or Baseline, or unwilling to refrain from use of recreational drugs during the study
26. Hypersensitivity to lemborexant or zolpidem or to their excipients
27. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5× the half-life, whichever is longer preceding informed consent
28. Previously participated in any clinical trial of lemborexant

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (60):
  - Jasper Summit Research LLC, Jasper, Alabama
  - PACT, Glendale, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Carlsbad, California
  - Southern California Research, Fountain Valley, California
  - Pacific Sleep Medicine Services, Oceanside, California
  - Research Center of Southern California, Oceanside, California
  - Orange County Neuropsychiatric Research Center, LLC, Orange, California
  - SDS Clinical Trials, Inc., Orange, California
  - Artemis Institute For Clinical Research LLC, San Diego, California
  - Pacific Research Network Inc, San Diego, California
  - Artemis Institute For Clinical Research, San Marcos, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Empire Clinical Research, Upland, California
  - PAB Clinical Research, Brandon, Florida
  - Saint Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Fleming Island Center For Clinical Research, Fleming Island, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - MD Clinical, Hallandale, Florida
  - QPS MRA, Hollywood, Florida
  - Quest Pharmaceutical Services-Miami Research Associates, LLC (QPS MRA), Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Compass Research LLC, Orlando, Florida
  - NeuroMedical Research Institute, Panama City, Florida
  - Clinical Research Group of St Petersburg Inc, St. Petersburg, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - SleepCare Research Institute Inc, Stockbridge, Georgia
  - Northwestern University, Chicago, Illinois
  - Chicago Research Center Inc, Chicago, Illinois
  - Helene A Emsellem MD PC, Chevy Chase, Maryland
  - Sleep Disorders Center of the Mid-Atlantic, Glen Burnie, Maryland
  - Neurocare Inc, Newton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Novi, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - St. Louis Clinical Trials, St Louis, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - CLINiLABS, Inc., Eatontown, New Jersey
  - Winthrop University Hospital, Garden City, New York
  - Clinical Research Unit, New York, New York
  - University of Rochester, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Sleep Medicine Centers of Western New York, West Seneca, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Cleveland Sleep Research Center, Middleburg Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Sleepmed of South Carolina, Columbia, South Carolina
  - Pioneer Research Solutions, Houston, Texas
  - Sleep Disorders Center of the Mid-Atlantic, Vienna, Virginia
  - Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Canada (8):
  - Sleep and Fatigue Institute, Calgary, Alberta
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Markham, Ontario
  - Somni Research Inc., Markham, Ontario
  - Tri Hospital Sleep West, Mississauga, Ontario
  - Sleep Wake Disorders Clinic, Scarborough Village, Ontario
  - Toronto, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
- France (5):
  - Centre Hospitalier Universitaire de Bordeaux, Hopital Pellegrin, Bordeaux
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon Bourgogne, Dijon
  - Hôtel Dieu de Paris Hospital, Paris
  - Hopital Civil, Strasbourg
- Germany (8):
  - Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Advanced Sleep Research GmbH, Berlin
  - Emovis GmbH, Berlin
  - Studienzentrum Wilhelmshöhe, Kassel
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Somni Bene Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Italy (7):
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - ASST di Pavia - Fondazione Istituto Neurologico Mondino IRCCS, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Spain (10):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital San Rafael, A Coruña
  - Hospital Clinic de Barcelona, Badalona
  - Barcelona
  - Clinica del Son Estivill, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Instituto de Investigaciones del Sueño, Madrid
  - Hospital Universitario Araba - Txagorritxu, Vitoria-Gasteiz
- United Kingdom (4):
  - Papworth Hospital, Cambridge, Cambridge Shire
  - University of Surrey, Guildford, Surrey
  - Guys Hospital, London
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Kushida CA, Zammit GK, Cheng JY, Kumar D, Moline M. Effect of lemborexant on sleep architecture in participants with insomnia disorder and mild obstructive sleep apnea. Sleep Med. 2025 Mar;127:170-177. doi: 10.1016/j.sleep.2024.12.023. Epub 2024 Dec 17. PMID 39879708
- [Derived] Gotfried MH, Auerbach SH, Dang-Vu TT, Mishima K, Kumar D, Moline M, Malhotra M. Efficacy and safety of insomnia treatment with lemborexant in older adults: analyses from three clinical trials. Drugs Aging. 2024 Sep;41(9):741-752. doi: 10.1007/s40266-024-01135-8. Epub 2024 Aug 9. PMID 39120786
- [Derived] Citrome L, Juday TR, Lundwall C. Lemborexant and Daridorexant for the Treatment of Insomnia: An Indirect Comparison Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Oct 2;84(6):23m14851. doi: 10.4088/JCP.23m14851. PMID 37796657
- [Derived] Inoue Y, Nishida M, Kubota N, Koebis M, Taninaga T, Muramoto K, Ishikawa K, Moline M. Comparison of the treatment effectiveness between lemborexant and zolpidem tartrate extended-release for insomnia disorder subtypes defined based on polysomnographic findings. J Clin Sleep Med. 2023 Mar 1;19(3):519-528. doi: 10.5664/jcsm.10378. PMID 36472134
- [Derived] Chepke C, Jain R, Rosenberg R, Moline M, Yardley J, Pinner K, Kumar D, Perdomo C, Filippov G, Atkins N, Malhotra M. Improvement in fatigue and sleep measures with the dual orexin receptor antagonist lemborexant in adults with insomnia disorder. Postgrad Med. 2022 Apr;134(3):316-325. doi: 10.1080/00325481.2022.2049553. Epub 2022 Mar 20. PMID 35254948
- [Derived] Citrome L, Juday T, Frech F, Atkins N Jr. Lemborexant for the Treatment of Insomnia: Direct and Indirect Comparisons With Other Hypnotics Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2021 Jun 1;82:20m13795. doi: 10.4088/JCP.20m13795. PMID 34077032
- [Derived] Moline M, Zammit G, Cheng JY, Perdomo C, Kumar D, Mayleben D. Comparison of the effect of lemborexant with placebo and zolpidem tartrate extended release on sleep architecture in older adults with insomnia disorder. J Clin Sleep Med. 2021 Jun 1;17(6):1167-1174. doi: 10.5664/jcsm.9150. PMID 33590823
- [Derived] Rosenberg R, Murphy P, Zammit G, Mayleben D, Kumar D, Dhadda S, Filippov G, LoPresti A, Moline M. Comparison of Lemborexant With Placebo and Zolpidem Tartrate Extended Release for the Treatment of Older Adults With Insomnia Disorder: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1918254. doi: 10.1001/jamanetworkopen.2019.18254. PMID 31880796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 67 investigative sites in the United States, Spain, Germany, Canada, United Kingdom, and Italy from 31 May 2016 to 30 January 2018.
Pre-assignment Details: A total of 3537 participants were screened, of which 1006 participants were randomized to the treatment period. All participants who were subsequently randomized completed a Run-in Period before randomization to treatment period.
Groups:
- Placebo: Participants received lemborexant-matched placebo and zolpidem matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment Period.
- Zolpidem Tartrate Extended Release 6.25 mg: Participants received zolpidem tartrate extended release (ZOL ER) 6.25 milligram (mg) and lemborexant-matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment period.
- Lemborexant 5 mg: Participants received lemborexant 5 mg and zolpidem-matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment Period.
- Lemborexant 10 mg: Participants received lemborexant 10 mg and zolpidem-matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment Period.
Period: Overall Study
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Started | 208 | 263 | 266 | 269
Completed | 198 | 246 | 258 | 260
Not Completed | 10 | 17 | 8 | 9
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 6 | 2 | 3
Not completed — Other | 1 | 6 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 2
Not completed — Participant's choice | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.
Groups:
- Zolpidem Tartrate Extended Release 6.25 mg: Participants received zolpidem tartrate extended release (ZOL ER) 6.25 mg and lemborexant-matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg | Total
Number analyzed (Participants) | 208 | 263 | 266 | 269 | 1006
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (6.36) | 64.3 (7.12) | 63.7 (6.78) | 64.2 (6.88) | 63.9 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 226 | 229 | 230 | 869
  Male | 24 | 37 | 37 | 39 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 32 | 51 | 47 | 165
  Not Hispanic or Latino | 173 | 231 | 215 | 222 | 841
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 153 | 173 | 199 | 202 | 727
  Black or African American | 51 | 80 | 63 | 62 | 256
  Japanese | 1 | 1 | 0 | 0 | 2
  Chinese | 1 | 0 | 0 | 1 | 2
  Other Asian | 0 | 4 | 2 | 4 | 10
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific | 0 | 2 | 0 | 0 | 2
  Other | 2 | 3 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Latency to Persistent Sleep (LPS) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 29/30
Description: LPS is defined as the time in minutes from lights off to the first epoch of 20 consecutive epochs of non- wakefulness as measured by PSG. Change from baseline to average LPS on Day 29 and 30 was reported.
Time Frame: Baseline, Days 29/30
Population: FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement at given time points.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
minutes
  Baseline | 43.89 (33.596) | 44.86 (36.528) | 44.61 (32.986)
  Change at Days 29/30: number analyzed (Participants) | 200 | 260 | 260
  Change at Days 29/30 | -7.93 (31.946) | -19.53 (33.054) | -21.46 (32.436)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Test type: Superiority; p = 0.0003, MMRM — Based on mixed effect model repeated measurement (MMRM) model with log transformation of LPS and factors for age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effects, and the baseline LPS as a covariate; Least Squares Geometric Mean(LSGM) Ratio = 0.773, 95% CI 2-sided [0.672 to 0.889]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with log transformation of LPS and factors for age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effects, and the baseline LPS as a covariate; LSGM Ratio = 0.723, 95% CI 2-sided [0.628 to 0.832]

2. Secondary Outcome: Change From Baseline in Mean Sleep Efficiency (SE) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 29/30
Description: SE is defined as percentage of time spent in bed asleep, calculated as total sleep time (TST) divided by interval from lights off until lights on as measured by PSG, multiplied by 100. Change from baseline to average SE on Day 29 and 30 was reported.
Time Frame: Baseline, Days 29/30
Population: The FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement at given time points.
Measure: Mean (Standard Deviation); unit: Percentage of time in bed asleep
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
Percentage of time in bed asleep
  Baseline | 68.89 (9.639) | 68.36 (11.268) | 67.85 (10.849)
  Change at Days 29/30: number analyzed (Participants) | 200 | 260 | 260
  Change at Days 29/30 | 5.35 (9.897) | 12.93 (9.741) | 14.09 (10.514)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effect, and the baseline SE as a covariate; Least Squares Mean (LSM) Difference = 7.07, 95% CI 2-sided [5.61 to 8.54], Standard Error of Mean 0.746
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; LSM Difference = 8.03, 95% CI 2-sided [6.57 to 9.49], Standard Error of Mean 0.746

3. Secondary Outcome: Change From Baseline in Mean Wake After Sleep Onset (WASO) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 29/30
Description: WASO is defined as minutes of wake from the onset of persistent sleep until lights on as measured by PSG. Change from baseline to average WASO on Days 29 and 30 was reported.
Time Frame: Baseline, Days 29/30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
minutes
  Baseline | 111.75 (37.179) | 113.44 (38.953) | 114.83 (39.997)
  Change at Days 29/30: number analyzed (Participants) | 200 | 260 | 260
  Change at Days 29/30 | -18.58 (41.931) | -43.89 (39.264) | -46.43 (39.595)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effect, and the baseline WASO as a covariate; LSM Difference = -23.96, 95% CI 2-sided [-29.98 to -17.95], Standard Error of Mean 3.068
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM; LSM Difference = -25.35, 95% CI 2-sided [-31.36 to -19.34], Standard Error of Mean 3.067

4. Secondary Outcome: Change From Baseline in WASO in the Second Half of the Night (WASO2H) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER on Days 29/30
Description: WASO2H is defined as time in minutes of wake during the interval from 240 minutes after lights off until lights on as measured by PSG. Change from baseline to average WASO2H on Days 29 and 30 was reported.
Time Frame: Baseline, Days 29/30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 262 | 266 | 269
minutes
  Baseline | 78.04 (33.849) | 76.60 (32.903) | 76.88 (32.126)
  Change at Days 29/30: number analyzed (Participants) | 250 | 260 | 260
  Change at Days 29/30 | -21.42 (36.257) | -27.19 (33.047) | -28.84 (33.138)
Statistical Analysis 1: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; Test type: Superiority — Based on MMRM model with factors of age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effect, and the baseline WASO2H as a covariate; p = 0.0038, MMRM; LSM Difference = -6.65, 95% CI 2-sided [-11.15 to -2.15], Standard Error of Mean 2.298
Statistical Analysis 2: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0005, MMRM; LSM Difference = -8, 95% CI 2-sided [-12.53 to -3.47], Standard Error of Mean 2.309

5. Other Pre Specified Outcome: Change From Baseline in Mean Body Sway Upon Awakening in the Morning for Lemborexant 5 mg and Lemborexant 10 mg Compared to Zolpidem ER on Days 2/3
Description: Body sway is detected through a cable around the participant's waist by the ataxia meter. Body sway is measured in units of one-third degree of the angle of arc. For ease in reporting, these are called arbitrary units, with a higher number indicating more body sway (less postural stability). Change from baseline in mean body sway on Days 2 and 3 was reported.
Time Frame: Baseline, Days 2/3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: one-third degree of angle of arc
Arm/Group | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 239 | 245 | 243
one-third degree of angle of arc
  Baseline | 26.96 (26.502) | 26.40 (20.781) | 36.29 (197.282)
  Change at Days 2/3: number analyzed (Participants) | 234 | 237 | 234
  Change at Days 2/3 | 8.47 (69.894) | -0.82 (20.383) | -8.97 (146.679)
Statistical Analysis 1: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; Zolpidem Tartrate Extended Release 6.25 mg v Lemborexant 5 mg; Test type: Superiority; p = 0.0171, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 2/3), and treatment-by-visit interaction as fixed effect, and the baseline posture stability of body sway as a covariate; LSM Difference = -9.63, 95% CI 2-sided [-17.53 to -1.72], Standard Error of Mean 4.029
Statistical Analysis 2: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; Zolpidem Tartrate Extended Release 6.25 mg v Lemborexant 10 mg; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSM Difference = -10.74, 95% CI 2-sided [-18.67 to -2.81], Standard Error of Mean 4.04

6. Other Pre Specified Outcome: Change From Baseline in Mean LPS, WASO, and TST of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER on Days 1/2 and Days 29/30
Description: LPS is defined as the time in minutes from lights off to the first epoch of 20 consecutive epochs of non-wakefulness as measured by the PSG. WASO is defined as minutes of wake from the onset of persistent sleep until lights on as measured by PSG. TST is defined as the amount of sleep in minutes from LPS until terminal awakening as measured by PSG. Change from baseline to average LPS, WASO, and TST on Days 1 and 2, and Days 29 and 30 were reported.
Time Frame: Baseline, Days 1/2, and Days 29/30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 262 | 266 | 269
minutes
  LPS: Baseline | 44.52 (38.349) | 44.86 (36.528) | 44.61 (32.986)
  LPS: Change at Days 1/2 | -12.56 (32.506) | -16.59 (28.742) | -19.48 (31.809)
  LPS: Change at Days 29/30: number analyzed (Participants) | 250 | 260 | 260
  LPS: Change at Days 29/30 | -7.51 (35.065) | -19.53 (33.054) | -21.46 (32.436)
  WASO: Baseline | 114.31 (39.992) | 113.44 (38.953) | 114.83 (39.997)
  WASO: Change at Days 1/2 | -44.36 (38.074) | -49.96 (39.578) | -59.59 (37.749)
  WASO: Change at Days 29/30: number analyzed (Participants) | 250 | 260 | 260
  WASO: Change at Days 29/30 | -36.50 (43.406) | -43.89 (39.264) | -46.43 (39.595)
  TST: Baseline | 326.99 (54.852) | 328.00 (54.224) | 325.07 (52.819)
  TST: Change at Days 1/2 | 55.31 (48.138) | 65.22 (46.695) | 79.58 (47.350)
  TST: Change at Days 29/30: number analyzed (Participants) | 250 | 260 | 260
  TST: Change at Days 29/30 | 43.34 (54.012) | 61.99 (46.817) | 67.86 (52.117)
Statistical Analysis 1: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; LPS, Days 1/2: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0218, MMRM — Based on MMRM model with log transformation of LPS and factors for age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline LPS as a covariate; LSGM Ratio = 0.874, 95% CI 2-sided [0.78 to 0.981]
Statistical Analysis 2: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; LPS, Days 1/2: Zolpidem ER, Lemborexant 10 mg; Test type: Other; p = 0.0006, MMRM — [p-value comment as in outcome 6, analysis 1]; LSGM Ratio = 0.818, 95% CI 2-sided [0.729 to 0.917]
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; LPS, Days 29/30: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LSGM Ratio = 0.634, 95% CI 2-sided [0.556 to 0.724]
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; LPS, Days 29/30: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; LSGM Ratio = 0.594, 95% CI 2-sided [0.521 to 0.677]
Statistical Analysis 5: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; WASO, Days 1/2: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0154, MMRM — Based on MMRM model with factors for age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline WASO as a covariate; LSM Difference = -6.16, 95% CI 2-sided [-11.15 to -1.17], Standard Error of Mean 2.544
Statistical Analysis 6: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; WASO, Days 1/2: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 6, analysis 5]; LSM Difference = -15.03, 95% CI 2-sided [-20.01 to -10.05], Standard Error of Mean 2.542
Statistical Analysis 7: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; WASO, Days 29/30: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0073, MMRM — Based on MMRM model with factors for age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effects, and the baseline WASO as a covariate; LSM Difference = -7.72, 95% CI 2-sided [-13.36 to -2.08], Standard Error of Mean 2.876
Statistical Analysis 8: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; WASO, Days 29/30: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0016, MMRM; LSM Difference = -9.1, 95% CI 2-sided [-14.75 to -3.45], Standard Error of Mean 2.883
Statistical Analysis 9: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; TST, Days 1/2: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.001, MMRM — Based on MMRM model with factors for age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline TST as a covariate; LSM Difference = 10.25, 95% CI 2-sided [4.18 to 16.32], Standard Error of Mean 3.094
Statistical Analysis 10: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; TST, Days 1/2: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 6, analysis 9]; LSM Difference = 23.1, 95% CI 2-sided [17.04 to 29.15], Standard Error of Mean 3.085
Statistical Analysis 11: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; TST, Days 29/30: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors for age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effects, and the baseline TST as a covariate; LSM Difference = 19.41, 95% CI 2-sided [12.63 to 26.2], Standard Error of Mean 3.457
Statistical Analysis 12: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; TST, Days 29/30: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 6, analysis 11]; LSM Difference = 24.1, 95% CI 2-sided [17.32 to 30.88], Standard Error of Mean 3.456

7. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Onset Latency (sSOL), Subjective Wake After Sleep Onset (sWASO) and Subjective Total Sleep Time (sTST) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER
Description: sSOL: estimated minutes from time attempted to sleep to sleep onset. sWASO: estimated minutes of wake at night after initial sleep onset to time stopped trying to sleep for the night. sTST: minutes of sleep from sleep onset to time stopped trying to sleep for the night. sSOL, sWASO, sTST were analyzed with diary handling rules (DHR) on an electronic sleep diary. Subjective measures were derived from sleep diaries entries, collected daily and analyzed at appropriate intervals.
Time Frame: First 7 nights (approximately Week 1) and Last 7 nights (approximately Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 259 | 264 | 269
minutes
  sSOL: Baseline: With DHR: number analyzed (Participants) | 258 | 263 | 269
  sSOL: Baseline: With DHR | 60.54 (36.350) | 65.79 (43.530) | 60.88 (42.514)
  sSOL: 1st 7 nights: With DHR: number analyzed (Participants) | 251 | 259 | 266
  sSOL: 1st 7 nights: With DHR | -16.23 (29.531) | -22.54 (32.812) | -21.88 (29.269)
  sSOL: last 7 nights: With DHR: number analyzed (Participants) | 246 | 252 | 258
  sSOL: last 7 nights: With DHR | -17.04 (30.683) | -25.20 (34.854) | -24.79 (34.068)
  sWASO: Baseline: With DHR: number analyzed (Participants) | 259 | 264 | 266
  sWASO: Baseline: With DHR | 173.06 (77.212) | 166.76 (82.047) | 175.35 (83.453)
  sWASO: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 253 | 261 | 262
  sWASO: Change at 1st 7 nights: With DHR | -48.91 (51.761) | -39.33 (55.022) | -55.06 (66.696)
  sWASO: Change at last 7 nights: With DHR: number analyzed (Participants) | 247 | 253 | 253
  sWASO: Change at last 7 nights: With DHR | -63.52 (64.161) | -44.51 (58.090) | -57.96 (72.791)
  sTST: Baseline: With DHR: number analyzed (Participants) | 247 | 253 | 258
  sTST: Baseline: With DHR | 273.07 (81.207) | 275.74 (83.650) | 266.10 (92.164)
  sTST: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 240 | 251 | 254
  sTST: Change at 1st 7 nights: With DHR | 56.99 (62.880) | 50.30 (60.065) | 67.80 (71.134)
  sTST: Change at last 7 nights: With DHR: number analyzed (Participants) | 235 | 245 | 244
  sTST: Change at last 7 nights: With DHR | 71.01 (76.574) | 62.41 (68.555) | 79.95 (81.211)
Statistical Analysis 1: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSOL, First 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0122, MMRM — Based on MMRM model model with log transformation of sSOL and factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSOL as a covariate; LSGM Ratio = 0.898, 95% CI 2-sided [0.825 to 0.977]
Statistical Analysis 2: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSOL, First 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 1]; LSGM Ratio = 0.83, 95% CI 2-sided [0.763 to 0.902]
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSOL, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0176, MMRM — Based on MMRM model model with log transformation of sSOL and factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSOL as a covariate; LSGM Ratio = 0.882, 95% CI 2-sided [0.796 to 0.978]
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSOL, Last 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model model with log transformation of sSOL and with factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSOL as a covariate; LSGM Ratio = 0.811, 95% CI 2-sided [0.732 to 0.899]
Statistical Analysis 5: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sWASO, First 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0706, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sWASO as a covariate; LSM Difference = 8.12, 95% CI 2-sided [-0.68 to 16.91], Standard Error of Mean 4.484
Statistical Analysis 6: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sWASO, First 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.1949, MMRM — [p-value comment as in outcome 7, analysis 5]; LSM Difference = -5.81, 95% CI 2-sided [-14.61 to 2.98], Standard Error of Mean 4.481
Statistical Analysis 7: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sWASO, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0059, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sWASO as a covariate; LSM Difference = 14.45, 95% CI 2-sided [4.16 to 24.73], Standard Error of Mean 5.241
Statistical Analysis 8: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sWASO, Last 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.3064, MMRM — [p-value comment as in outcome 7, analysis 7]; LSM Difference = 5.36, 95% CI 2-sided [-4.92 to 15.65], Standard Error of Mean 5.241
Statistical Analysis 9: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sTST, First 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.2174, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baselines sTST as a covariate; LSM Difference = -6.57, 95% CI 2-sided [-17.02 to 3.88], Standard Error of Mean 5.325
Statistical Analysis 10: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sTST, First 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0949, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sTST as a covariate; LSM Difference = 8.88, 95% CI 2-sided [-1.55 to 19.31], Standard Error of Mean 5.313
Statistical Analysis 11: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sTST, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.2718, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sTST as a covariate; LSM Difference = -6.82, 95% CI 2-sided [-19.01 to 5.36], Standard Error of Mean 6.207
Statistical Analysis 12: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sTST, Last 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.2317, MMRM — [p-value comment as in outcome 7, analysis 11]; LSM Difference = 7.43, 95% CI 2-sided [-4.75 to 19.61], Standard Error of Mean 6.206

8. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Efficiency (sSE) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER
Description: sSE: percentage of sTST per subjective time spent in bed asleep, calculated as the interval from the time attempted to sleep to time stopped trying to sleep for the night, and time spent asleep derived from subjective time spent in bed minus sWASO. sWASO: estimated minutes of wake at night after initial sleep onset to time stopped trying to sleep for the night. sSE was analyzed with DHR on an electronic sleep diary. Subjective measures were derived from sleep diaries entries, collected daily and analyzed at appropriate intervals.
Time Frame: First 7 nights (approximately Week 1) and Last 7 nights (approximately Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of subjective time in bed asleep
Groups:
- Zolpidem Tartrate Extended Release 6.25 mg: Participants received ZOL ER 6.25 mg and lemborexant-matched placebo, tablets, orally, once daily from Day 1 up to Day 30 in the Treatment period.
Arm/Group | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 247 | 253 | 258
% of subjective time in bed asleep
  sSE: Baseline: With DHR | 55.49 (15.802) | 56.05 (17.094) | 54.31 (18.318)
  sSE: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 240 | 251 | 254
  sSE: Change at 1st 7 nights: With DHR | 11.96 (12.526) | 10.56 (12.296) | 13.97 (14.188)
  sSE: Change at last 7 nights: With DHR: number analyzed (Participants) | 235 | 245 | 244
  sSE: Change at last 7 nights: With DHR | 14.83 (15.011) | 12.92 (13.884) | 16.12 (16.300)
Statistical Analysis 1: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSE, First 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.1963, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSE as a covariate; LSM Difference = -1.37, 95% CI 2-sided [-3.46 to 0.71], Standard Error of Mean 1.063
Statistical Analysis 2: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSE, First 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSE as a covariate; p = 0.1093, MMRM; LSM Difference = 1.7, 95% CI 2-sided [-0.38 to 3.78], Standard Error of Mean 1.06
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSE, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.2196, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSE as a covariate; LSM Difference = -1.53, 95% CI 2-sided [-3.98 to 0.92], Standard Error of Mean 1.247
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSE, Last 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.4013, MMRM — [p-value comment as in outcome 8, analysis 3]; LSM Difference = 1.05, 95% CI 2-sided [-1.4 to 3.49], Standard Error of Mean 1.246

9. Other Pre Specified Outcome: Change From Baseline in Mean LPS, WASO, WASO2H, and TST of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 1/2
Description: LPS: amount of time in minutes from lights off to first epoch of 20 consecutive epochs of non-wakefulness. WASO: amount of time in minutes of wake from the onset of persistent sleep until lights. WASO2H: amount of time in minutes of wake during the interval from 240 minutes after lights off until lights on. TST: amount of time in minutes of sleep from sleep onset until terminal awakening. LPS, WASO, WASO2H, and TST were measured by PSG. Change from baseline to average LPS, WASO, WASO2H, and TST on Day 1 and 2 were reported.
Time Frame: Baseline, Days 1/2
Population: FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
minutes
  LPS: Baseline | 43.89 (33.596) | 44.86 (36.528) | 44.61 (32.986)
  LPS: Change at Days 1/2 | -6.45 (32.618) | -16.59 (28.742) | -19.48 (31.809)
  WASO: Baseline | 111.75 (37.179) | 113.44 (38.953) | 114.83 (39.997)
  WASO: Change at Days 1/2 | -15.07 (36.938) | -49.96 (39.578) | -59.59 (37.749)
  WASO2H: Baseline | 74.44 (30.109) | 76.60 (32.903) | 76.88 (32.126)
  WASO2H: Change at Days 1/2 | -7.06 (31.097) | -30.28 (32.056) | -37.10 (30.815)
  TST: Baseline | 330.67 (46.268) | 328.00 (54.224) | 325.07 (52.819)
  TST: Change at Days 1/2 | 19.44 (43.348) | 65.22 (46.695) | 79.58 (47.350)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; LPS: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0092, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline LPS as a covariate; LSGM Ratio = 0.85, 95% CI 2-sided [0.752 to 0.961]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; LPS: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0002, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days1/2), and treatment-by-visit interaction as fixed effects, and the baseline LPS as a covariate; LSGM Ratio = 0.795, 95% CI 2-sided [0.704 to 0.899]
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; WASO: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effect, and the baseline WASO as a covariate; LSM Difference = -33.4, 95% CI 2-sided [-38.71 to -28.09], Standard Error of Mean 2.711
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; WASO: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 9, analysis 3]; LSM Difference = -42.27, 95% CI 2-sided [-47.57 to -36.97], Standard Error of Mean 2.705
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; WASO2H: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline WASO2H as a covariate; LSM Difference = -21.66, 95% CI 2-sided [-26.01 to -17.3], Standard Error of Mean 2.221
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; WASO2H: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 9, analysis 5]; LSM Difference = -28.33, 95% CI 2-sided [-32.68 to -23.98], Standard Error of Mean 2.219
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; TST: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effect, and the baseline TST as a covariate; LSM Difference = 44.05, 95% CI 2-sided [37.59 to 50.51], Standard Error of Mean 3.291
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; TST: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 9, analysis 7]; LSM Difference = 56.9, 95% CI 2-sided [50.46 to 63.34], Standard Error of Mean 3.284

10. Other Pre Specified Outcome: Change From Baseline in Mean SE of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 1/2
Description: SE is defined as percentage of time spent in bed asleep, calculated as TST divided by interval from lights off until lights on as measured by PSG, multiplied by 100. Change from baseline to average SE on Day 1 and 2 were reported.
Time Frame: Baseline, Days 1/2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of time in bed asleep
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
Percentage of time in bed asleep
  SE: Baseline | 68.89 (9.639) | 68.36 (11.268) | 67.85 (10.849)
  SE: Change at Days 1/2 | 4.22 (9.033) | 13.60 (9.725) | 16.48 (9.623)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; SE: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effects, and the baseline SE as a covariate; LSM Difference = 9.01, 95% CI 2-sided [7.7 to 10.31], Standard Error of Mean 0.666
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; SE: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 1/2), and treatment-by-visit interaction as fixed effect, and the baseline SE as a covariate; LSM Difference = 11.6, 95% CI 2-sided [10.3 to 12.9], Standard Error of Mean 0.664

11. Other Pre Specified Outcome: Change From Baseline in Mean WASO2H and TST of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo on Days 29/30
Description: WASO2H is defined as the time in minutes of wake during the interval from 240 minutes after lights off until lights on. TST is defined as the amount of sleep in minutes from sleep onset until terminal awakening. WASO and TST were measured by PSG. Change from baseline to average WASO and TST on Day 29 and 30 were reported.
Time Frame: Baseline, Days 29/30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 266 | 269
minutes
  WASO2H: Baseline | 74.44 (30.109) | 76.60 (32.903) | 76.88 (32.126)
  WASO2H: Days 29 /30: number analyzed (Participants) | 200 | 260 | 260
  WASO2H: Days 29 /30 | -8.92 (31.909) | -27.19 (33.047) | -28.84 (33.138)
  TST: Baseline | 330.67 (46.268) | 328.00 (54.224) | 325.07 (52.819)
  TST: Days 29/30: number analyzed (Participants) | 200 | 260 | 260
  TST: Days 29/30 | 25.65 (47.587) | 61.99 (46.817) | 67.86 (52.117)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; WASO2H: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effect, and the baseline WASO2H as a covariate; LSM Difference = -16.41, 95% CI 2-sided [-21.23 to -11.6], Standard Error of Mean 2.457
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; WASO2H: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 1]; LSM Difference = -17.76, 95% CI 2-sided [-22.57 to -12.96], Standard Error of Mean 2.451
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; TST: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 29/30), and treatment-by-visit interaction as fixed effect, and the baseline TST as a covariate; LSM Difference = 34.16, 95% CI 2-sided [26.95 to 41.36], Standard Error of Mean 3.673
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; TST: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 3]; LSM Difference = 38.85, 95% CI 2-sided [31.64 to 46.05], Standard Error of Mean 3.672

12. Other Pre Specified Outcome: Change From Baseline in Mean sSOL, sWASO, and sTST of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo
Description: sSOL: estimated minutes from time attempted to sleep to sleep onset. sWASO: estimated minutes of wake at night after initial sleep onset to time stopped trying to sleep for the night. sTST: minutes of sleep from sleep onset to time stopped trying to sleep for the night. sSOL, sWASO, sTST were analyzed with DHR on an electronic sleep diary. Subjective measures were derived from sleep diaries entries, collected daily and analyzed at appropriate intervals.
Time Frame: First 7 nights (approximately Week 1) and Last 7 nights (approximately Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 206 | 264 | 269
minutes
  sSOL: Baseline: With DHR: number analyzed (Participants) | 206 | 263 | 269
  sSOL: Baseline: With DHR | 55.90 (37.389) | 65.79 (43.530) | 60.88 (42.514)
  sSOL: Change at 1st 7 nights :With DHR: number analyzed (Participants) | 202 | 259 | 266
  sSOL: Change at 1st 7 nights :With DHR | -6.83 (23.040) | -22.54 (32.812) | -21.88 (29.269)
  sSOL: Change at last 7 nights: With DHR: number analyzed (Participants) | 196 | 252 | 258
  sSOL: Change at last 7 nights: With DHR | -8.10 (27.447) | -25.20 (34.854) | -24.79 (34.068)
  sWASO: Baseline: With DHR: number analyzed (Participants) | 206 | 264 | 266
  sWASO: Baseline: With DHR | 170.89 (80.676) | 166.76 (82.047) | 175.35 (83.453)
  sWASO: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 202 | 261 | 262
  sWASO: Change at 1st 7 nights: With DHR | -27.92 (45.201) | -39.33 (55.022) | -55.06 (66.696)
  sWASO: Change at last 7 nights: With DHR: number analyzed (Participants) | 196 | 253 | 253
  sWASO: Change at last 7 nights: With DHR | -36.01 (57.584) | -44.51 (58.090) | -57.96 (72.791)
  sTST: Baseline: With DHR: number analyzed (Participants) | 201 | 253 | 258
  sTST: Baseline: With DHR | 276.23 (87.649) | 275.74 (83.650) | 266.10 (92.164)
  sTST: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 197 | 251 | 254
  sTST: Change at 1st 7 nights: With DHR | 30.86 (57.437) | 50.30 (60.065) | 67.80 (71.134)
  sTST: Change at last 7 nights: With DHR: number analyzed (Participants) | 190 | 245 | 244
  sTST: Change at last 7 nights: With DHR | 38.98 (66.174) | 62.41 (68.555) | 79.95 (81.211)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; sSOL, First 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (First 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSOL as a covariate; LSGM Ratio = 0.815, 95% CI 2-sided [0.745 to 0.891]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; sSOL, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 12, analysis 1]; LSGM Ratio = 0.753, 95% CI 2-sided [0.689 to 0.823]
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; sSOL, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Last 7 Nights), and treatment-by-visit interaction as fixed effects, and the baseline sSOL as a covariate; LSGM Ratio = 0.75, 95% CI 2-sided [0.671 to 0.837]
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; sSOL, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 12, analysis 3]; LSGM Ratio = 0.689, 95% CI 2-sided [0.618 to 0.769]
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; sWASO, First 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0093, MMRM — [p-value comment as in outcome 7, analysis 5]; LSM Difference = -12.41, 95% CI 2-sided [-21.76 to -3.06], Standard Error of Mean 4.764
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; sWASO, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 5]; LSM Difference = -26.34, 95% CI 2-sided [-35.68 to -16.99], Standard Error of Mean 4.762
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; sWASO, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0396, MMRM — [p-value comment as in outcome 7, analysis 7]; LSM Difference = -11.49, 95% CI 2-sided [-22.42 to -0.55], Standard Error of Mean 5.573
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; sWASO, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 7, analysis 7]; LSM Difference = -20.57, 95% CI 2-sided [-31.51 to -9.63], Standard Error of Mean 5.574
Statistical Analysis 9: Comparison: Placebo vs Lemborexant 5 mg; sTST, First 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 7, analysis 9]; LSM Difference = 19.05, 95% CI 2-sided [8.03 to 30.08], Standard Error of Mean 5.619
Statistical Analysis 10: Comparison: Placebo vs Lemborexant 10 mg; sTST, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 9]; LSM Difference = 34.51, 95% CI 2-sided [23.5 to 45.52], Standard Error of Mean 5.609
Statistical Analysis 11: Comparison: Placebo vs Lemborexant 5 mg; sTST, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 7, analysis 11]; LSM Difference = 23.57, 95% CI 2-sided [10.68 to 36.45], Standard Error of Mean 6.565
Statistical Analysis 12: Comparison: Placebo vs Lemborexant 10 mg; sTST, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 7, analysis 11]; LSM Difference = 37.82, 95% CI 2-sided [24.94 to 50.71], Standard Error of Mean 6.565

13. Other Pre Specified Outcome: Change From Baseline in Mean sSE of Lemborexant 10 mg and Lemborexant 5 mg Compared to Placebo
Description: as for outcome 8
Time Frame: First 7 nights (approximately Week 1) and Last 7 nights (approximately Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of subjective time in bed asleep
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 201 | 253 | 258
% of subjective time in bed asleep
  sSE: Baseline: With DHR | 56.08 (17.343) | 56.05 (17.094) | 54.31 (18.318)
  sSE: Change at 1st 7 nights: With DHR: number analyzed (Participants) | 197 | 251 | 254
  sSE: Change at 1st 7 nights: With DHR | 6.73 (10.930) | 10.56 (12.296) | 13.97 (14.188)
  sSE: Change at last 7 nights: With DHR: number analyzed (Participants) | 190 | 245 | 244
  sSE: Change at last 7 nights: With DHR | 8.35 (13.273) | 12.92 (13.884) | 16.12 (16.300)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; sSE, First 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 8, analysis 1]; LSM Difference = 3.76, 95% CI 2-sided [1.56 to 5.97], Standard Error of Mean 1.122
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; sSE, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 1]; LSM Difference = 6.84, 95% CI 2-sided [4.64 to 9.04], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; sSE, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 8, analysis 3]; LSM Difference = 4.61, 95% CI 2-sided [2.02 to 7.19], Standard Error of Mean 1.319
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; sSE, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 8, analysis 3]; LSM Difference = 7.18, 95% CI 2-sided [4.6 to 9.77], Standard Error of Mean 1.319

14. Other Pre Specified Outcome: Percentage of Responders With Objective and Subjective Sleep Onset Response, and Objective and Subjective Sleep Maintenance Response
Description: Objective sleep onset response: LPS less than or equal to (<=) 20 minutes (mins) provided baseline LPS was greater than (>) 30 mins. Subjective sleep onset response: sSOL <=20 mins provided mean baseline sSOL was >30 mins. Objective sleep maintenance response: WASO <=60 minutes provided baseline WASO was >60 mins and was reduced by >10 mins compared to baseline. Subjective sleep maintenance response: sWASO <=60 mins provided mean WASO was >60 mins and was reduced by >10 mins compared to baseline. Subjective measures were derived from sleep diaries entries, collected daily and analyzed at appropriate intervals. Average data for Days 1 and 2, Days 29 and 30, and first and last 7 nights of treatment period was reported.
Time Frame: Days 1/2, Days 29/30, first 7 night (approximately Week 1), and Last seven nights (approximately Week 4)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 263 | 266 | 269
percentage of participants
  LPS: Days 1/2 | 15.4 | 10.3 | 15.8 | 17.8
  LPS: Days 29/30 | 15.9 | 11.4 | 20.3 | 22.3
  sSOL: First 7 nights (with DHR) | 2.9 | 7.6 | 9.8 | 10.4
  sSOL: Last 7 nights (with DHR) | 7.2 | 8.7 | 16.9 | 14.5
  WASO: Days 1/2 | 16.8 | 46.0 | 51.1 | 64.3
  WASO: Days 29/30 | 22.1 | 34.6 | 44.4 | 46.1
  sWASO: First 7 nights (with DHR) | 9.6 | 16.7 | 16.9 | 20.4
  sWASO: Last 7 nights (with DHR) | 15.4 | 23.2 | 23.3 | 23.0
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; LPS, Days 1/2: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.9028, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 0.41, 95% CI 2-sided [-6.22 to 7.04]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; LPS, Days 1/2: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.4699, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 2.49, 95% CI 2-sided [-4.2 to 9.18]
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; LPS, Days 1/2: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0566, Cochran-Mantel-Haenszel; Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 5.58, 95% CI 2-sided [-0.14 to 11.31]
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; LPS, Days 1/2: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0122, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.57, 95% CI 2-sided [1.71 to 13.44]
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; LPS, Days 29/30: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.2176, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 4.42, 95% CI 2-sided [-2.5 to 11.34]
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; LPS, Days 29/30: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0773, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 6.47, 95% CI 2-sided [-0.55 to 13.49]
Statistical Analysis 7: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; LPS, Days 29/30: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 8.85, 95% CI 2-sided [2.68 to 15.02]
Statistical Analysis 8: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; LPS, Days 29/30: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 10.89, 95% CI 2-sided [4.61 to 17.17]
Statistical Analysis 9: Comparison: Placebo vs Lemborexant 5 mg; sSOL, First 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 6.9, 95% CI 2-sided [2.66 to 11.14]
Statistical Analysis 10: Comparison: Placebo vs Lemborexant 10 mg; sSOL, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.5, 95% CI 2-sided [3.19 to 11.81]
Statistical Analysis 11: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSOL, First 7 nights: Zolpidem, Lemborexant 5 mg; Test type: Superiority; p = 0.3643, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 2.22, 95% CI 2-sided [-2.56 to 7.01]
Statistical Analysis 12: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSOL, First 7 nights: Zolpidem, Lemborexant 10 mg; Test type: Superiority; p = 0.2553, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 2.82, 95% CI 2-sided [-2.02 to 7.66]
Statistical Analysis 13: Comparison: Placebo vs Lemborexant 5 mg; sSOL, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 9.69, 95% CI 2-sided [3.98 to 15.4]
Statistical Analysis 14: Comparison: Placebo vs Lemborexant 10 mg; sSOL, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0128, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.29, 95% CI 2-sided [1.8 to 12.79]
Statistical Analysis 15: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sSOL, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0051, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 8.16, 95% CI 2-sided [2.51 to 13.81]
Statistical Analysis 16: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sSOL, Last 7nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0389, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 5.76, 95% CI 2-sided [0.34 to 11.18]
Statistical Analysis 17: Comparison: Placebo vs Lemborexant 5 mg; WASO, Days 1/2: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 34.26, 95% CI 2-sided [26.46 to 42.06]
Statistical Analysis 18: Comparison: Placebo vs Lemborexant 10 mg; WASO, Days 1/2: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 47.57, 95% CI 2-sided [40.02 to 55.13]
Statistical Analysis 19: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; WASO, Days 1/2: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.2534, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 4.89, 95% CI 2-sided [-3.49 to 13.28]
Statistical Analysis 20: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; WASO: Days 1/2: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 18.25, 95% CI 2-sided [10.1 to 26.4]
Statistical Analysis 21: Comparison: Placebo vs Lemborexant 5 mg; WASO, Days 29/30: Placebo, Lemborexant 5 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 22.2, 95% CI 2-sided [14.06 to 30.35]
Statistical Analysis 22: Comparison: Placebo vs Lemborexant 10 mg; WASO, Days 29/30: Placebo, Lemborexant 10 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 24.13, 95% CI 2-sided [16.16 to 32.1]
Statistical Analysis 23: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; WASO, Days 29/30: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 9.59, 95% CI 2-sided [1.36 to 17.81]
Statistical Analysis 24: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; WASO, Days 29/30: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0058, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 11.43, 95% CI 2-sided [3.38 to 19.48]
Statistical Analysis 25: Comparison: Placebo vs Lemborexant 5 mg; sWASO, First 7 nights: Placebo, Lemborexant 5; Test type: Superiority; p = 0.0222, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.3, 95% CI 2-sided [1.27 to 13.33]
Statistical Analysis 26: Comparison: Placebo vs Lemborexant 10 mg; sWASO, First 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 10.84, 95% CI 2-sided [4.57 to 17.11]
Statistical Analysis 27: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sWASO, First 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.9495, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 0.21, 95% CI 2-sided [-6.17 to 6.58]
Statistical Analysis 28: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sWASO: First 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.2708, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 3.72, 95% CI 2-sided [-2.88 to 10.32]
Statistical Analysis 29: Comparison: Placebo vs Lemborexant 5 mg; sWASO, Last 7 nights: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0322, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.91, 95% CI 2-sided [0.86 to 14.96]
Statistical Analysis 30: Comparison: Placebo vs Lemborexant 10 mg; sWASO, Last 7 nights: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0363, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 7.69, 95% CI 2-sided [0.68 to 14.71]
Statistical Analysis 31: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; sWASO, Last 7 nights: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.9885, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = 0.05, 95% CI 2-sided [-7.14 to 7.24]
Statistical Analysis 32: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; sWASO, Last 7 nights: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.9651, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by age group; Difference of Percentage = -0.16, 95% CI 2-sided [-7.31 to 6.99]

15. Other Pre Specified Outcome: Change From Baseline in Score From Items 4 to 7 on the Insomnia Severity Index (ISI) of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER and Placebo on Day 31
Description: The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated were: severity of sleep onset; sleep maintenance; early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of the sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale was used to rate each item (from 0 = no problem to 4 = very severe problem) yielding a total score from 0 to 28.
Time Frame: Baseline and Day 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 263 | 266 | 269
score on scale
  Baseline | 11.21 (2.436) | 11.06 (2.508) | 10.91 (2.419) | 10.84 (2.334)
  Change at Day 31: number analyzed (Participants) | 198 | 244 | 257 | 253
  Change at Day 31 | -3.88 (3.559) | -5.24 (3.764) | -4.83 (3.593) | -4.77 (3.735)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0006, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = -1.1, 95% CI 2-sided [-1.73 to -0.47], Standard Error of Mean 0.319
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0007, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = -1.08, 95% CI 2-sided [-1.71 to -0.46], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.2951, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = 0.32, 95% CI 2-sided [-0.28 to 0.91], Standard Error of Mean 0.301
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.2744, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = 0.33, 95% CI 2-sided [-0.26 to 0.92], Standard Error of Mean 0.303

16. Other Pre Specified Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Score of Lemborexant 10 mg and Lemborexant 5 mg Compared to Zolpidem ER and Placebo on Day 31
Description: The FSS is a self-report scale on which participants are instructed to choose a number from 1 to 7 that indicates their degree of agreement with each of 9 statements about their fatigue where "1" indicates strongly disagree, and "7" indicates strongly agree. The FSS total score was the sum of all responses to the 9 questions. The FSS average item score was the average of the score for each item. Higher total scores and higher average item scores indicated greater fatigue.
Time Frame: Baseline and Day 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 263 | 266 | 269
score on scale
  Baseline | 37.48 (13.602) | 37.15 (13.788) | 37.47 (13.518) | 37.42 (13.111)
  Change at Day 31 | -6.75 (11.916) | -7.80 (12.879) | -8.14 (13.411) | -8.00 (14.058)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.2348, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline FSS as a covariate; LSM Difference = -1.26, 95% CI 2-sided [-3.35 to 0.82], Standard Error of Mean 1.063
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.2745, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline FSS as a covariate; LSM Difference = -1.17, 95% CI 2-sided [-3.26 to 0.93], Standard Error of Mean 1.067
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.711, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = -0.37, 95% CI 2-sided [-2.35 to 1.6], Standard Error of Mean 1.005
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.7854, ANCOVA — Based on ANCOVA model with factors of age group, region, treatment and the baseline ISI as a covariate; LSM Difference = -0.27, 95% CI 2-sided [-2.26 to 1.71], Standard Error of Mean 1.009

17. Other Pre Specified Outcome: Change From Baseline in Mean Power of Attention (POA) and Speed of Memory Retrieval (SOMT) on Days 2/3
Description: POA reflects the ability to focus attention and process information. POA is calculated from the sum of simple reaction time, choice reaction time and digit vigilance. SOMT reflects time taken to retrieve information from working and episodic memory. SOMT is a composite score created by combining numerical working memory and spatial working memory and word recognition and picture recognition. Cognitive performance assessment was done by a computerized performance assessment battery (PAB) which was administered on a laptop computer. A positive change from baseline reflects impairment and a lower value of decrease from baseline indicates better performance. Change from baseline to average POA and SOMT on Days 2 and 3 was reported.
Time Frame: Baseline, Days 2/3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 208 | 263 | 266 | 269
millisecond
  POA: Baseine: number analyzed (Participants) | 195 | 239 | 249 | 246
  POA: Baseine | 1421.0 (210.27) | 1418.7 (195.95) | 1452.9 (263.04) | 1399.2 (192.47)
  POA : Days 2/3: number analyzed (Participants) | 186 | 233 | 240 | 236
  POA : Days 2/3 | -14.2 (149.31) | 37.1 (107.15) | 8.9 (154.33) | 31.1 (142.38)
  SOMT: Baseline: number analyzed (Participants) | 195 | 238 | 246 | 246
  SOMT: Baseline | 4507.7 (1098.73) | 4513.8 (1097.65) | 4674.3 (1174.74) | 4619.8 (1065.00)
  SOMT: Days 2/3: number analyzed (Participants) | 186 | 232 | 237 | 235
  SOMT: Days 2/3 | -177.9 (668.77) | 60.7 (749.12) | -185.1 (645.18) | -152.8 (722.49)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; POA: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.0141, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 2/3), and treatment-by-visit interaction as fixed effects, and the baseline POA as a covariate; LSM Difference = 30.77, 95% CI 2-sided [6.23 to 55.31], Standard Error of Mean 12.505
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; POA: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.0016, MMRM — [p-value comment as in outcome 17, analysis 1]; LSM Difference = 39.67, 95% CI 2-sided [15.05 to 64.29], Standard Error of Mean 12.542
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; POA: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.1031, MMRM — [p-value comment as in outcome 17, analysis 1]; LSM Difference = -19.22, 95% CI 2-sided [-42.34 to 3.9], Standard Error of Mean 11.779
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; POA: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.3825, MMRM — [p-value comment as in outcome 17, analysis 1]; LSM Difference = -10.32, 95% CI 2-sided [-33.5 to 12.86], Standard Error of Mean 11.813
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; SOMT: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.6348, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 2/3), and treatment-by-visit interaction as fixed effects, and the baseline SOMT as a covariate; LSM Difference = 28.81, 95% CI 2-sided [-90.18 to 147.8], Standard Error of Mean 60.626
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; SOMT: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.4026, MMRM — [p-value comment as in outcome 17, analysis 5]; LSM Difference = 50.83, 95% CI 2-sided [-68.3 to 169.97], Standard Error of Mean 60.702
Statistical Analysis 7: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; SOMT: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 17, analysis 5]; LSM Difference = -203.36, 95% CI 2-sided [-315.56 to -91.15], Standard Error of Mean 57.171
Statistical Analysis 8: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; SOMT: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0016, MMRM — [p-value comment as in outcome 17, analysis 5]; LSM Difference = -181.33, 95% CI 2-sided [-293.71 to -68.96], Standard Error of Mean 57.255

18. Other Pre Specified Outcome: Change From Baseline in Mean Quality of Memory (QOM) and Continuity of Attention (COA) on Days 2/3
Description: QOM represents the ability to store information in memory and subsequently retrieve it. It is a composite score created by combining accuracy measures from 2 sets of working memory and 4 sets of episodic memory. Two sets of working memory were included: numerical and spatial working memory, and ranges from -2 to 2. Four sets of episodic memory were included: immediate and delayed word recall, and word and picture recognition, and ranges from -200 to 400. COA is the ability to sustain attention. Number of correct responses (out of 50) for choice reaction time was added to total number of targets correctly identified (out of 45) digit vigilance minus number of false alarms (total score of -45 to 95). Higher values were better. Change from baseline to average QOM and COA on Days 2 and 3 was reported.
Time Frame: Baseline, Days 2/3
Population: FAS was group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose efficacy measurement at given time points.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 195 | 239 | 249 | 246
units on scale
  QOM: Baseline: number analyzed (Participants) | 195 | 239 | 248 | 246
  QOM: Baseline | 342.2 (66.03) | 350.0 (65.30) | 345.7 (67.60) | 340.7 (72.75)
  QOM: Change at Days 2/3: number analyzed (Participants) | 185 | 233 | 239 | 235
  QOM: Change at Days 2/3 | 3.5 (45.20) | -12.1 (46.94) | 1.4 (44.21) | -2.8 (44.11)
  COA: Baseline | 90.7 (4.77) | 90.6 (6.0) | 91.0 (5.15) | 91.3 (4.15)
  COA: Change at Days2/3: number analyzed (Participants) | 186 | 233 | 240 | 236
  COA: Change at Days2/3 | 0.0 (4.16) | -1.0 (4.48) | 0.2 (4.95) | -0.7 (3.92)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; QOM: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.9936, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 2/3), and treatment-by-visit interaction as fixed effects, and the baseline QOM as a covariate; LSM Difference = -0.03, 95% CI 2-sided [-8.16 to 8.09], Standard Error of Mean 4.141
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; QOM: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.1595, MMRM — [p-value comment as in outcome 18, analysis 1]; LSM Difference = -5.85, 95% CI 2-sided [-14 to 2.3], Standard Error of Mean 4.154
Statistical Analysis 3: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; QOM: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 18, analysis 1]; LSM Difference = 12.73, 95% CI 2-sided [5.09 to 20.38], Standard Error of Mean 3.894
Statistical Analysis 4: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; QOM: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.0774, MMRM — [p-value comment as in outcome 18, analysis 1]; LSM Difference = 6.92, 95% CI 2-sided [-0.76 to 14.6], Standard Error of Mean 3.913
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; COA: Placebo, Lemborexant 5 mg; Test type: Superiority; p = 0.3726, MMRM — Based on MMRM model with factors of age group, region, treatment, visit (Days 2/3), and treatment-by-visit interaction as fixed effects, and the baseline COA as a covariate; LSM Difference = 0.35, 95% CI 2-sided [-0.42 to 1.12], Standard Error of Mean 0.393
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; COA: Placebo, Lemborexant 10 mg; Test type: Superiority; p = 0.2579, MMRM — [p-value comment as in outcome 18, analysis 5]; LSM Difference = -0.45, 95% CI 2-sided [-1.22 to 0.33], Standard Error of Mean 0.394
Statistical Analysis 7: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 5 mg; COA: Zolpidem ER, Lemborexant 5 mg; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 18, analysis 5]; LSM Difference = 1.39, 95% CI 2-sided [0.66 to 2.11], Standard Error of Mean 0.37
Statistical Analysis 8: Comparison: Zolpidem Tartrate Extended Release 6.25 mg vs Lemborexant 10 mg; COA: Zolpidem ER, Lemborexant 10 mg; Test type: Superiority; p = 0.112, MMRM — [p-value comment as in outcome 18, analysis 5]; LSM Difference = 0.59, 95% CI 2-sided [-0.14 to 1.32], Standard Error of Mean 0.372

ADVERSE EVENTS:
Time Frame: Run-in Phase (Day -7) up to End of treatment (Day 44)
Groups:
- Run -in Period Placebo: Participants received lemborexant-matched placebo and zolpidem matched placebo, tablets, orally, once on each night for 7 consecutive nights up to Baseline (Day 1), immediately before the time the participant intended to try to sleep of run-in period.
Arm/Group | Placebo | Zolpidem Tartrate Extended Release 6.25 mg | Lemborexant 5 mg | Lemborexant 10 mg | Run -in Period Placebo
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/263 | 0/266 | 0/268 | 0/1006
Serious Adverse Events (participants affected / at risk) | 0/209 | 4/263 | 2/266 | 0/268 | 0/1006
Other Adverse Events (participants affected / at risk) | 16/209 | 18/263 | 27/266 | 28/268 | 34/1006
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=209) | Zolpidem Tartrate Extended Release 6.25 mg (N=263) | Lemborexant 5 mg (N=266) | Lemborexant 10 mg (N=268) | Run -in Period Placebo (N=1006)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=209) | Zolpidem Tartrate Extended Release 6.25 mg (N=263) | Lemborexant 5 mg (N=266) | Lemborexant 10 mg (N=268) | Run -in Period Placebo (N=1006)
Headache (Nervous system disorders) | 13 (13) | 14 (21) | 17 (21) | 13 (15) | 34 (34)
Somnolence (Nervous system disorders) | 4 (4) | 4 (5) | 11 (11) | 19 (20) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT02783729/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT02783729/SAP_001.pdf